CLINICAL TRIAL: NCT00422292
Title: An Immunogenicity, Safety, and Non-Interference Evaluation of Pediatric Vaccines Administered Concomitantly With Menactra® (Meningococcal [Groups A, C, Y and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) to Healthy Toddlers
Brief Title: Immunogenicity and Safety of Pediatric Vaccines When Administered With Menactra® in Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTA37
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Meningitis; Measles; Mumps; Rubella; Varicella
Keywords: Menactra vaccine; Meningococcal meningitis; Measles; Mumps; Rubella; Varicella vaccines; Haemophilus influenzae type b; Pneumococcal conjugate vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Measles; Mumps; Rubella; Chickenpox; Haemophilus Infections | interventions — Meningococcal Vaccines; measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Menactra® at 9 and 12 Months (Experimental): Participants will received Menactra® vaccination at 9 and 12 months of age.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine
- Menactra® at 9 Months and Menactra® + MMRV at 12 Months (Experimental): Participants will receive Menactra® at 9 months of age and Menactra® plus measles, mumps, rubella, varicella (MMRV) vaccine at 12 months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine
- Menactra® at 9 Months and Menactra® + PCV at 12 Months (Experimental): Participants will receive Menactra® at 9 months of age and Menactra® plus pneumococcal conjugate vaccine (PCV) at 12 months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine
- MMRV + PCV at 12 Months (Active Comparator): Participants who received no vaccination at 9 months of age and measles, mumps, rubella, varicella (MMRV) vaccine plus pneumococcal conjugate vaccine (PCV) at 12 months of age
  Interventions: Biological: Measles, Mumps, Rubella and Varicella

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL dose, intramuscular (IM)
  Other Names: Menactra®
  Arms: Menactra® at 9 and 12 Months
Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL dose, IM
  Other Names: Menactra®
  Arms: Menactra® at 9 Months and Menactra® + MMRV at 12 Months
Biological: Meningococcal Polysaccharide Diphtheria Conjugate Vaccine — 0.5 Ml dose, IM
  Other Names: Menactra®
  Arms: Menactra® at 9 Months and Menactra® + PCV at 12 Months
Biological: Measles, Mumps, Rubella and Varicella — 0.5 mL dose, SC
  Other Names: ProQuad®; M-M-R®II
  Arms: MMRV + PCV at 12 Months

SUMMARY:
This is a modified single-blind, randomized, parallel-group, comparative, multicenter study to test Menactra vaccine in toddlers.

Primary Objectives:

* To evaluate the antibody responses induced by Measles, Mumps, Rubella, and Varicella (MMRV) vaccine when administered alone or concomitantly with Menactra vaccine.
* To evaluate the antibody responses induced by Pneumococcal Conjugated Vaccine (PCV) when administered alone or concomitantly with Menactra vaccine.

Observational Objectives:

Safety - To describe the safety profile throughout the course of the study from Day 0 up to 6 months after the last study vaccination[s]) in subjects in the study groups.

Immunogenicity:

- To describe the antibody responses to meningococcal serogroups A, C, Y, and W-135, 30 days after the first and second Menactra vaccine administration in a subset of subjects in the first study group.

DETAILED DESCRIPTION:
No meningococcal vaccine is presently licensed for the population aged < 2 years in the US, establishing the effectiveness of a quadrivalent polysaccharide conjugate vaccine against invasive meningococcal disease in children aged < 2 years would address this important, currently unmet public health need.

At enrollment, each 9-month old subject will be randomly assigned to a study group and vaccinated. A second vaccination will be administered at 12 months of age. Subjects will provide one blood sample during the trial.

Twelve-month old subjects will also be vaccinated with routine pediatric vaccines and provide one blood sample 30 days after vaccinations in the control group

ELIGIBILITY:
Inclusion Criteria :

* Healthy, as determined by medical history and physical examination
* Aged 9 months (249 to 291 days) for Groups 1, 2, and 3 or aged 12 months (365 to 386 days) for Group 4 at the time of enrollment
* The parent or legal guardian has signed and dated the Institutional Review Board (IRB)-approved informed consent form.

Exclusion Criteria :

* Serious acute or chronic disease (e.g., cardiac, renal, metabolic, rheumatologic, psychiatric, hematologic, autoimmune disorders, diabetes, atopic conditions, congenital defects, convulsions, encephalopathy, blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic system, acute untreated tuberculosis) that could interfere with trial conduct or completion
* Known or suspected impairment of immunologic function
* Acute medical illness within the last 72 hours or a temperature ≥ 100.4ºF (≥38.0ºC) at the time of enrollment.
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C seropositivity as reported by the parent or legal guardian
* Received either immune globulin or other blood products within the last 3 months, or received injected or oral corticosteroids, or other immunomodulator therapy within 6 weeks of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting < 7 days and individuals (e.g., asthmatics) on a short schedule of oral steroids lasting 3 to 4 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment. Topical steroids are not included in this exclusion criterion.
* Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to any blood draw. Topical antibiotics and antibiotic drops are not included in this exclusion criterion.
* Suspected or known hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the study vaccines or a vaccine containing the same substances. For ProQuad vaccine recipients, this includes a hypersensitivity to gelatin or a history of anaphylactic reactions to neomycin.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination.
* Parent or legal guardian unable or unwilling to comply with the study procedures
* Participation in another interventional clinical trial in the 30 days preceding enrollment or planned participation in another clinical trial involving the investigation of a drug, vaccine, medical procedure, or medical device during the subject's trial period.
* Diagnosed with any condition, which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine
* Received any vaccine in the 30-day period prior to receipt of the study vaccines, or scheduled to receive any vaccination other than influenza vaccination and hyposensitization therapy in the 30-day period after receipt of the study vaccines. Hyposensitization therapy and influenza vaccination may be received up to two weeks before or two weeks after receiving the study vaccines. Subjects should not have received their fourth dose of Pneumococcal conjugate vaccine (PCV) or Haemophilus influenzae type b (Hib) vaccine or their first dose of Measles, mumps, rubella, varicella (MMRV) vaccine before enrollment or been scheduled to receive these vaccines outside of the study-specified visits.
* Personal or family history of Guillain-Barré Syndrome (GBS)
* History of seizures, including febrile seizures, or any other neurologic disorder
* Known hypersensitivity to dry natural rubber latex.

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1664 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (78):
- United States (77):
  - Tuscaloosa, Alabama
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Atascadero, California
  - Fresno, California
  - Paramount, California
  - Roseville, California
  - Sacramento, California
  - San Jose, California
  - Torrance, California
  - Aurora, Colorado
  - Norwich, Connecticut
  - Viera, Florida
  - West Palm Beach, Florida
  - Dalton, Georgia
  - Marietta, Georgia
  - Tifton, Georgia
  - Woodstock, Georgia
  - Chicago, Illinois
  - Fishers, Indiana
  - Dubuque, Iowa
  - Owensboro, Kentucky
  - Bossier City, Louisiana
  - Perry Hall, Maryland
  - Woburn, Massachusetts
  - Niles, Michigan
  - Stevensville, Michigan
  - Bridgeton, Missouri
  - Kansas City, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Bellevue, Nebraska
  - La Vista, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Whitehouse Station, New Jersey
  - Brooklyn, New York
  - Fishkill, New York
  - Hopewell Junction, New York
  - Ithaca, New York
  - Lake Success, New York
  - Mineola, New York
  - New York, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - Boone, North Carolina
  - Clyde, North Carolina
  - Durham, North Carolina
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Independence, Ohio
  - Strongsville, Ohio
  - Harleysville, Pennsylvania
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Wexford, Pennsylvania
  - Clarksville, Tennessee
  - Kingsport, Tennessee
  - Houston, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Lehi, Utah
  - Ogden, Utah
  - Pleasant Grove, Utah
  - Provo, Utah
  - South Jordan, Utah
  - Springville, Utah
  - St. George, Utah
  - Urem, Utah
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
  - Huntington, West Virginia
  - Morgantown, West Virginia
  - Marshfield, Wisconsin
- San Juan, PR, Puerto Rico

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 January 2007 to 16 March 2008 in 92 clinical centers in the US.
Pre-assignment Details: A total of 2289 participants who met the inclusion and exclusion criteria were enrolled and vaccinated; 1643 were included in the final analyses presented.
  625 participants that got ActHIB as part of their 12 month study vaccinations prior to Protocol Amendment 2 approval were excluded from all analyses and presented in a separate report.
Groups:
- Group 1: Menactra® at 9 and 12 Months: Participants who received only Menactra® vaccination at 9 and 12 months of age
- Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months: Participants who received Menactra® at 9 months of age and Menactra® plus measles, mumps, rubella, varicella (MMRV or MMR+V) vaccine at 12 months of age
- Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months: Participants who received Menactra® at 9 months of age and Menactra® plus pneumococcal conjugate vaccine (PCV) at 12 months of age
- Group 4: MMRV + PCV at 12 Months: Participants who received no vaccination at 9 months of age and measles, mumps, rubella, varicella (MMRV) vaccine plus pneumococcal conjugate vaccine (PCV) at 12 months of age
Period: Overall Study
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Started | 257 | 664 | 246 | 476
Completed | 239 | 598 | 224 | 452
Not Completed | 18 | 66 | 22 | 24
Not completed — Serious adverse events | 1 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 4 | 25 | 8 | 5
Not completed — Lost to Follow-up | 6 | 12 | 6 | 6
Not completed — Withdrawal by Subject | 6 | 25 | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months | Total
Number analyzed (Participants) | 257 | 664 | 246 | 476 | 1643
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 257 | 664 | 246 | 476 | 1643
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 283.4 (11.3) | 283.0 (11.3) | 282.8 (10.3) | 374.8 (8.6) | 283.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 349 | 118 | 231 | 817
  Male | 138 | 315 | 128 | 245 | 826
Region of Enrollment [Number; unit: participants]
  United States | 257 | 664 | 246 | 476 | 1643

OUTCOME MEASURES:

1. Primary Outcome: Measles, Mumps, Rubella, and Varicella (MMRV) Antibody Values in Participants Who Received MMRV Vaccine (Groups 2 and 4 Only)
Description: Percentage of participants who had a concentration of ≥ 300 mIU/mL in the enzyme-linked immunosorbent assay (ELISA) or ≥ 120 mIU/mL in the neutralization when the ELISA concentration was less than 300 mIU/mL - for measles; ≥ 500 U/mL (ELISA) or ≥ 60 (1/dil) in the neutralization assay when the ELISA concentration was less than 500 mIU/mL - for mumps; ≥ 10 IU/mL (ELISA) - for Rubella; and ≥ 300 mIU/mL (ELISA) or ≥ 4 (1/dil) Fluorescent antibody to membrane antigen (FAMA) when the ELISA concentration was less than 300 mIU/mL - for varicella.
Time Frame: Day 30 after the 12-month vaccination
Population: Antibody responses were evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Number analyzed (Participants) | 0 | 498 | 0 | 399
Percentage of Participants
  Measles |  | 98 |  | 98
  Mumps |  | 95 |  | 95
  Rubella |  | 93 |  | 88
  Varicella |  | 93 |  | 87

2. Primary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Pneumococcal Antibodies After Pneumococcal Conjugated Vaccine (PCV) in Groups 3 and 4
Time Frame: Day 30 after the 12-month vaccination
Population: Geometric Mean Concentrations (GMCs) were determined in the per-protocol population Group 3 and Group 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Number analyzed (Participants) | 0 | 0 | 191 | 399
Titers
  Serotype 4 |  |  | 1.82 [1.62 to 2.05] | 3.33 [3.06 to 3.62]
  Serotype 6B |  |  | 5.40 [4.79 to 6.09] | 10.8 [9.89 to 11.7]
  Serotype 9V |  |  | 2.06 [1.84 to 2.30] | 3.57 [3.29 to 3.88]
  Serotype 14 |  |  | 6.73 [5.95 to 7.60] | 10.5 [9.65 to 11.3]
  Serotype 18C |  |  | 1.58 [1.43 to 1.75] | 2.91 [2.66 to 3.18]
  Serotype 19F |  |  | 2.50 [2.24 to 2.78] | 4.03 [3.74 to 4.34]
  Serotype 23F |  |  | 4.62 [4.06 to 5.25] | 7.03 [6.39 to 7.73]

3. Other Pre Specified Outcome: Percentage of Participants With Anti-Pneumococcal Concentrations ≥ 0.35 μg/mL After Pneumococcal Conjugate Vaccine (PCV) in Group 3 and Group 4
Time Frame: Day 30 after 12-month vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Number analyzed (Participants) | 0 | 0 | 191 | 399
Percentage of Participants
  Serotype 4 |  |  | 98 | 99
  Serotype 6B |  |  | 100 | 100
  Serotype 9V |  |  | 100 | 100
  Serotype 14 |  |  | 100 | 100
  Serotype18C |  |  | 98 | 99
  Serotype 19F |  |  | 100 | 100
  Serotype 23F |  |  | 100 | 100

4. Other Pre Specified Outcome: Percentage of Participants Reporting a Solicited Injection Site and Systemic Reactions After Menactra® Vaccination at 9 Months of Age
Description: Solicited injection site reactions: Injection site tenderness, injection site erythema, and injection site swelling.
  Solicited systemic reactions: Fever (temperature), vomiting, crying abnormal, drowsiness, appetite lost, and irritability.
Time Frame: Days 0 to 7 after vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Number analyzed (Participants) | 257 | 616 | 246 | 0
Percentage of Participants
  Any Solicited Injection Site Reacton | 46 | 43 | 49 |
  Any Tenderness | 35 | 33 | 38 |
  Grade 3 Tenderness (Cries when limb is moved) | 0 | 1 | 0 |
  Any Erythema | 23 | 20 | 23 |
  Grade 3 Erythema (≥ 2.0 in) | 2 | 1 | 2 |
  Any Swelling | 13 | 11 | 9 |
  Grade 3 Swelling (≥ 2.0 in) | 1 | 0 | 0 |
  Any Solicited Systemic Reaction | 66 | 69 | 71 |
  Any Fever | 10 | 13 | 13 |
  Grade 3 Fever (> 103.1 ºF or > 39.5 ºC) | 0 | 1 | 1 |
  Any Vomiting | 17 | 12 | 15 |
  Grade 3 Vomiting | 1 | 1 | 0 |
  Any Crying Abnormal | 37 | 34 | 34 |
  Grade 3 Crying Abnormal (> 3 hours) | 3 | 3 | 2 |
  Any Irritability | 56 | 56 | 51 |
  Grade 3 Irritability (Inconsolable) | 5 | 3 | 2 |
  Any Drowsiness | 33 | 32 | 35 |
  Grade 3 Drowsiness (Sleeps most of time) | 1 | 1 | 0 |
  Any Appetite Lost | 26 | 26 | 26 |
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 1 | 2 | 0 |

5. Other Pre Specified Outcome: Percentage of Participants With Solicited Injection Site and Systemic Reactions After Vaccination at 12 Months of Age
Time Frame: Days 0 to 7 after vaccination
Population: Solicited Injection Site and Systemic Reactions were assessed in the intend-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Months | Group 3: Menactra® at 9 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Number analyzed (Participants) | 257 | 572 | 246 | 476
Percentage of Participants
  Any Solicited Injection Site Reaction - Menactra | 44 | 46 | 57 | 0
  Any Tenderness | 34 | 38 | 51 | 0
  Grade 3 Tenderness (Cries when limb is moved) | 0 | 1 | 1 | 0
  Any Erythema | 24 | 23 | 27 | 0
  Grade 3 Erythema (≥ 2.0 in) | 3 | 3 | 3 | 0
  Any Swelling | 13 | 13 | 15 | 0
  Grade 3 Swelling (≥ 2.0 in) | 1 | 1 | 1 | 0
  Any Solicited Injection Site Reaction - MMRV | 0 | 38 | 0 | 49
  Any Tenderness | 0 | 32 | 0 | 42
  Grade 3 Tenderness (Cries when limb is moved) | 0 | 1 | 0 | 0
  Any Erythema | 0 | 18 | 0 | 23
  Grade 3 Erythema (≥ 2.0 in) | 0 | 2 | 0 | 1
  Any Swelling | 0 | 11 | 0 | 12
  Grade 3 Swelling (≥ 2.0 in) | 0 | 1 | 0 | 0
  Any Solicited Injection Site Reaction - PCV | 0 | 0 | 54 | 62
  Any Tenderness | 0 | 0 | 49 | 52
  Grade 3 Tenderness (Cries when limb is moved) | 0 | 0 | 0 | 0
  Any Erythema | 0 | 0 | 28 | 34
  Grade 3 Erythema (≥ 2.0 in) | 0 | 0 | 3 | 3
  Any Swelling | 0 | 0 | 17 | 22
  Grade 3 Swelling (≥ 2.0 in) | 0 | 0 | 1 | 2
  Any Solicited Systemic Reaction | 56 | 70 | 69 | 77
  Any Fever | 10 | 21 | 16 | 24
  Grade 3 Fever (> 103.1 ºF or > 39.5 ºC) | 0 | 3 | 3 | 3
  Any Vomiting | 7 | 10 | 7 | 10
  Grade 3 Vomiting | 0 | 1 | 0 | 0
  Any Crying Abnormal | 22 | 41 | 35 | 39
  Grade 3 Crying Abnormal (> 3 hours) | 1 | 3 | 2 | 2
  Any Irritability | 43 | 58 | 60 | 62
  Grade 3 Irritability (Inconsolable) | 4 | 4 | 4 | 4
  Any Drowsiness | 25 | 32 | 34 | 39
  Grade 3 Drowsiness (Sleeps most of time) | 0 | 1 | 1 | 2
  Any Appetite Lost | 24 | 32 | 27 | 29
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 1 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 6 months after the last vaccination.
Groups:
- Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Month: Participants who received Menactra® at 9 months of age and Menactra® plus measles, mumps, rubella, varicella (MMRV or MMR+V) vaccine at 12 months of age
- Group 3: Menactra® at 12 Months; Menactra® + PCV at 12 Months: Participants who received Menactra® at 9 months of age and Menactra® plus pneumococcal conjugate vaccine (PCV) at 12 months of age
Arm/Group | Group 1: Menactra® at 9 and 12 Months | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Month | Group 3: Menactra® at 12 Months; Menactra® + PCV at 12 Months | Group 4: MMRV + PCV at 12 Months
Serious Adverse Events (participants affected / at risk) | 14/257 | 24/616 | 10/246 | 17/476
Other Adverse Events (participants affected / at risk) | 91/257 | 185/664 | 77/246 | 148/476
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® at 9 and 12 Months (N=257) | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Month (N=616) | Group 3: Menactra® at 12 Months; Menactra® + PCV at 12 Months (N=246) | Group 4: MMRV + PCV at 12 Months (N=476)
Congenital spinal cord anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected Cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kawasaki's diseas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Closed head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniosynostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (3) | 6 (6) | 1 (1) | 4 (4)
Myoclonic epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® at 9 and 12 Months (N=257) | Group 2: Menactra® at 9 Months; Menactra® + MMRV at 12 Month (N=664) | Group 3: Menactra® at 12 Months; Menactra® + PCV at 12 Months (N=246) | Group 4: MMRV + PCV at 12 Months (N=476)
Diarrhoea (Gastrointestinal disorders) | 18 (21) | 38 (42) | 12 (12) | 29 (33)
Teething (Gastrointestinal disorders) | 13 (16) | 27 (32) | 17 (20) | 15 (17)
Pyrexia (General disorders) | 10 (10) | 14 (15) | 2 (2) | 48 (51)
Nasopharyngitis (Infections and infestations) | 13 (13) | 18 (18) | 7 (7) | 10 (11)
Otitis media (Infections and infestations) | 24 (25) | 52 (52) | 22 (22) | 20 (20)
Upper respiratory tract infection (Infections and infestations) | 22 (22) | 50 (51) | 25 (26) | 19 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 28 (29) | 6 (7) | 16 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 25 (27) | 8 (8) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications